CLINICAL TRIAL: NCT03975543
Title: Natural History Study of Retinitis Pigmentosa in Patient Carrying Pathogenic Mutations in RHO, PDE6A or PDE6B.
Brief Title: Retrospective Natural History Study of Retinitis Pigmentosa
Acronym: PHENOROD1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: SparingVision (Industry)
Responsible Party: Sponsor
Other Study IDs: PHENOROD1
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Retinitis Pigmentosa (RP)
Keywords: Retinitis Pigmentosa; RHO; PDE6A; PDE6B; Pathogenic mutation; Retrospective; Natural History; Retinal Disease; Eye Diseases; Blindness; Inherited Eye Diseases; Vision Disorders; Inherited Retinal Disorders; Rod-Cone Dystrophy
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Eye Diseases; Blindness; Vision Disorders; Cone-Rod Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is natural history study of rods and cones degenerations in patients with Retinitis Pigmentosa (RP) caused by pathogenic mutations in RHO, PDE6A or PDE6B gene mutations.

DETAILED DESCRIPTION:
This is a retrospective, longitudinal, observational case history study to determine the natural history of rods and cones degeneration in patients diagnosed with RP caused by pathogenic mutations in genes with selective expression in rods: rhodopsin (RHO), phosphodiesterase 6A (PDE6A) or phosphodiesterase 6B (PDE6B).

113 participants will be enrolled in this study at the single center: CHNO-CIC Quinze-Vingt Paris in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RP caused by pathogenic mutations in RHO, PDE6A or PDE6B genes.

Exclusion Criteria:

* Patients with a pathogenic mutation in any other gene known to be involved in RP.
* Patients with any ocular disorder other than RP, likely to impact the retinal function.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with RP caused by pathogenic mutations in RHO, PDE6A or PDE6B gene mutations.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 2 years
  Progression of disease over time as measured by best corrected visual acuity (BCVA) (ETDRS, Snellen) and refraction
Visual field | 2 years
  Progression of disease over time as measured by visual fields (kinetic and static)
Spectral Domain Optical Coherence tomography (SD-OCT) | 2 years
  Progression of disease over time as measured by SD-OCT (EZ length, ELM length, ONL thickness, macular volume).
Fundus Autofluorescence (FAF) | 2 years
  Progression of disease as measured by FAF (Hyperautofluorescent ring)

SECONDARY OUTCOMES:
Patients characteristics | 2 years
  Age, gender, medical and surgical history, family history and concomitant treatments
Clinical diagnosis | baseline (At diagnosis)
  Age and description at onset, clinical signs, relevant treatments and an ophthalmological anamnesis
Genetic diagnosis | baseline (At diagnosis)
  Mutated gene, identified pathogenic mutation
Electroretinogram (ERG) | baseline (At diagnosis)
  Photopic and scotopic full field
Color vision | 2 years
  15 Hue Desaturated Lanthony

CONTACTS AND LOCATIONS:
Locations (1):
- CHNO XV-XX Paris - CIC 1423, Paris, France